CLINICAL TRIAL: NCT01541150
Title: Neuropsychological Approach of Pedophilic Behaviors, a Pilot Study in a Population of Inmates Pedophilic Offenders
Brief Title: Impaired Decision Making in Pedophilic Offenders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8673; 2011-A00402-39 (Other: ID-RCB)
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2012-02

CONDITIONS: Pedophilia
Keywords: Pedophilia; Impaired Decision making; Insight; Cognitive Distorsions; Impulsiveness
MeSH Terms: conditions — Pedophilia; Impulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient suffering pedophilia (Active Comparator): This group is the active comparator because patients suffering pedophilia with neuropsychological questionnaires
  Interventions: Behavioral: neuropsychological questionnaires
- control group (Placebo Comparator): This group is the placebo comparator
  Interventions: Behavioral: neuropsychological questionnaires

INTERVENTIONS:
Behavioral: neuropsychological questionnaires — Due to this study population (inmates), the investigators have decided to classify the protocol as and interventionnal study.

SUMMARY:
Pedophilic behaviors represent a public health problem with serious consequences. The investigators hypothesize a disruption in the decision-making strategies among sex offenders pedophiles. Highlight this type of abnormality would offer a specific treatment of a possible neuropsychological deficit (with cognitive remediation for instance) and perhaps avoid recurrences of this type of behavior.

DETAILED DESCRIPTION:
Cross-sectional study, comparing a group of 64 pedophilic offenders inmates condamned with a group of 64 volunteers non-pedophiles matched by age and level of study.

ELIGIBILITY:
Inclusion Criteria:

* For the controls, lack of diagnosis of disorders of sexual behavior (paraphilias) current or past (DSM IV)
* For the pedophilic offenders:

  * Placement and conviction for rape or sexual assault of a minor under 15 years
  * Recognition of the facts
  * Existence of a current or past diagnosis of pedophilia (according to the DSM IV).

Exclusion Criteria:

* Presence of a current major depressive episode (DSM IV - MINI)
* History of cerebral neurological disorder or a cranial trauma with loss of consciousness current
* IGT test already done
* Schizophrenia or Other current psychotic disorders(according to the criteria DSM IV of MINI test).
* taking psychoactive drug

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-08 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of neuropsychological performances between control group and group of persons suffering from pedophilia | 36 months (at the end of the study)
  Bring to light cognitive changes in the pedophilia, by comparing the neuropsychological performances of a group of persons suffering from pedophilia to a control group (no pedophile).
  The neuropsychological performances between two groups are assessed by neuropsychologic questionnaires (Iowa Gambling Task, MINI 5.0.0, MADRS, Test de Rolls, N-Back, WAIS III, go-no-go...)

CONTACTS AND LOCATIONS:
Overall Officials: Lacambre Mathieu, MD, Principal Investigator — CHU de Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, France